CLINICAL TRIAL: NCT05875311
Title: Usefulness of a Telemonitoring System to Optimize Continuity of Care From Cardiology to Primary Care in Patients With Chronic Coronary Syndrome
Brief Title: Telemonitoring System for Improving Continuity of Care in Patients With Chronic Coronary Syndrome (TELSINCORC)
Acronym: TELSINCORC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catcronic Salut SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TRISA-2023
Record Dates: First submitted 2023-03-18; First posted 2023-05-25 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Chronic Coronary Syndrome
Keywords: mobile health; Chronic coronary syndrome; cardiac rehabilitation; telerehabilitation; secondary prevention; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Pragmatic, open-label, prospective, parallel-group study
Who Masked: Outcomes Assessor
Masking Description: The characteristics of the interventions do not allow the study to be blinded either for the patient or for the professional. However, the analyses and surveys will be performed in a masked manner without the assigned group being identified by the investigators who carry out the examinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemonitoring (Experimental): Patients in the intervention group will come to the ambulatory centre 2 times, undergoing mobile application training and the same educational talks as in the control group. Subsequently, they will follow the scheduled physical activities and adherence to the risk factor management according to individualised guidelines in their App, until the end of the study period. All data generated are recorded on the professional website. The degree of compliance with the objectives set is monitored by means of 7 coloured icons, which vary according to the target achievement.
  Interventions: Device: telemonitoring
- control follow-up (Other): Patients in the control group will come to the ambulatory centre only once. The same educational talks as to the intervention group will be given. A conventional outpatient follow-up by primary care and the corresponding specialist will be carried out.
  Interventions: Other: control follow-up

INTERVENTIONS:
Device: telemonitoring — The system consists of the following elements:
  Professional website at the ambulatory centre, which allows:
  To set up an individualised care plan To establish the patient's risk profile and targets for improvement. Long-term monitoring of the evolution of cardiovascular risk factors and events that occurred Advise the patient on self-management strategies.
  Mobile application software with the following functions:
  Scheduled exercise sessions Medication reminder Measurement reminder (weight, blood pressure, heart rate, waist circumference, etc.) Messages: Inbox folder for system messages and messages generated by professionals for a specific patient or video conference.
  Training monitor: guides the patient in the performance of their exercise. Access to certified health information for patients
  Arms: telemonitoring
Other: control follow-up — Patients are instructed to perform 150 minutes per week of moderate physical activity and follow healthy lifestyles
  Arms: control follow-up

SUMMARY:
In a randomized clinical trial, a comprehensive telerehabilitation system with a prolonged follow-up strategy demonstrated superiority over a control group with centre-based cardiac rehabilitation in terms of physical activity, VO2 max, adherence to a Mediterranean diet, lipid particle profile and cost-effectiveness. The aim of this study is to demonstrate an extension of the benefit to patients with chronic coronary syndrome in primary care.

DETAILED DESCRIPTION:
The patients who have suffered an acute coronary event have a recurrence rate of 2.5% to 15.5% person-years during the first year. Control of cardiovascular risk factors can improve the prognosis of these patients. Following the results of a clinical trial to validate a comprehensive monitoring system called Cardioplan, with a prolonged monitoring strategy, The investigators aim to conduct a study in patients with chronic coronary syndrome in the primary care setting comparing a control group with standard follow-up and a 10-month telemonitored group. Four primary care centres will participate. Two health centres attend mainly a population with a medium-high upper socioeconomic level and the other two mainly a population with a medium-low socioeconomic level. A total of 160 subjects are expected to be included in the follow-up, with 80 subjects in each study group. The primary endpoint is to demonstrate that telemonitored follow-up improves functional exercise capacity compared to usual care, by assessing the distance in meters covered in the 6-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients after more than one year of an acute coronary syndrome of both sexes.
* Age equal to or less than 72 years.

Exclusion Criteria:

* Refusal of informed consent
* Advanced biological age.
* Kidney failure (GFR < 30ml/min/1.73 m2).
* Liver failure (GOT >2 times normal value).
* Ejection fraction less than 50%.
* Uncontrolled blood pressure (>140/90 mmHg).
* Uncontrolled heart failure.
* Dissecting aortic aneurysm.
* Uncontrolled ventricular tachycardia or other dangerous ventricular arrhythmias.
* Aortic or mitral valve disease.
* Recent systemic or pulmonary embolism.
* Active or recent thrombophlebitis.
* Acute infectious diseases.
* Uncontrolled supraventricular arrhythmias or tachycardia.
* Repeated or frequent ventricular ectopic activity.
* Moderate pulmonary hypertension.
* Ventricular aneurysm.
* Uncontrolled diabetes, thyrotoxicosis, myxedema,
* Conduction disorders such as: complete atrioventricular block. Left bundle branch block.
* Wolf-Parkinson-White syndrome.
* Fixed rate pacing.
* Severe anaemia.
* Psychoneurotic disorders.
* Neuromuscular, musculoskeletal and arthritic disorders that may limit activity. may limit activity.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The 6-min walk distance (6MWD) | 10 months
  Meters (m)

SECONDARY OUTCOMES:
Maximal heart rate in the six minute walk test | 10 months
  beats per minute (bpm)
Total cholesterol | 10 months
  mg/dL
Glycosylated haemoglobin | 10 months
  Percentage (%)
Weight | 10 months
  Kilograms (Kg)
Waist circumference | 10 months
  waist circumference change (cm)
Visceral fat | 10 months
  percentage (%)
Energy expenditure obtained from the International Physical Activity questionnaire (IPAQ) questionaire | 10 months
  Kcal/week
High level of effort obtained from the International Physical Activity questionnaire (IPAQ) questionaire | 10 months
  percentage
Total score of Adherence to Mediterranean Diet obtained from the Prevention with Mediterranean Diet questionnaire (PREDIMED). | 10 months
  Units. Minimum value: 0, maximum value: 14. Higher scores mean a better outcome.
Global score of emotional distress obtained from the Hospital Anxiety and Depression Scale (HADS) | 10 months
  Units. Minimum value: 0, maximum value: 14. Lower scores mean a better outcome.
Anxiety subscale of emotional distress obtained from the Hospital Anxiety and Depression Scale (HADS) | 10 months
  Units. Minimum value: 0, maximum value: 7. Lower scores mean a better outcome.
Depression subscale of Emotional distress obtained from the Hospital Anxiety and Depression Scale (HADS) | 10 months
  Units. Minimum value: 0, maximum value: 7. Lower scores mean a better outcome.
Global index of the health-related quality of life obtained from the European Quality of Life questionnaire (EuroQol-5D) | 10 months
  Units. Minimum value: 0, maximum value: 1. Higher scores mean a better outcome.
Health status obtained from the European Quality of Life questionnaire (EuroQol-5D) | 10 months
  Units. Minimum value: 0, maximum value: 100. Higher scores mean a better outcome.
smoking cessation | 10 months
  percentage
User's experience from the System Usability Scale (SUS) score | 10 months
  Units. Minimum value: 0, maximum value: 100. Higher scores mean a better outcome.
Cost-effectiveness analysis | 10 months
  net cost divided by changes in health outcomes
Body mass Index | 10 months
  weight and height will be combined to report BMI (kg/m^2)
High | 10 months
  centimeters (cm)
Percentage expected for age and sex in the six minute walk test | 10 months
  Percentage
Leukocyte count | 10 month
  WBCs per microliter
Neutrophil count | 10 monts
  Neutrophils per microliter and percentage of white blood cells
Lymphocyte count | 10 month
  Lymphocytes per microliter and percentage of white blood cells
Platelet count | 10 month
  Platelets per microliter
GlycA | 10 monts
  μmol/L
Small LDL particles | 10 months
  μmol/L
Physical activity derived from the International Physical Activity questionnaire (IPAQ) | 10 months
  self-reported physical activity measured in metabolic equivalents (MET-min/week) Minimum value: 0, maximum value 19,278. Higher scores mean a better outcome.
HDL cholesterol | 10 months
  mg/dL
LDL cholesterol | 10 months
  mg/dL
Non-HDL cholesterol | 10 months
  mg/dL
Triglycerides | 10 months
  mg/dL
Apolipoprotein B/Apolipoprotein A-I ratio | 10 months
  Units

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Dalli Peydró, MD, Principal Investigator — Hospital Arnau de VIlanova. Valencia
Locations (1):
- Hospital Arnau de Vilanova, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalli-Peydro E, Gisbert-Criado R, Amigo N, Sanz-Sevilla N, Cosin-Sales J. Cardiac telerehabilitation with long-term follow-up reduces GlycA and improves lipoprotein particle profile: A randomised controlled trial. Int J Cardiol. 2022 Dec 15;369:60-64. doi: 10.1016/j.ijcard.2022.08.017. Epub 2022 Aug 6. PMID 35944773
- [Background] Dalli Peydro E, Sanz Sevilla N, Tuzon Segarra MT, Miro Palau V, Sanchez Torrijos J, Cosin Sales J. A randomized controlled clinical trial of cardiac telerehabilitation with a prolonged mobile care monitoring strategy after an acute coronary syndrome. Clin Cardiol. 2022 Jan;45(1):31-41. doi: 10.1002/clc.23757. Epub 2021 Dec 24. PMID 34952989
- [Background] Paoli G, Notarangelo MF, Mattioli M, La Sala R, Foa C, Solinas E, Fusco S, Fava C, Caminiti C, Artioli G, Pela G, Dall'Aglio E, Manari A, Tondi S, Rizzo A, Trapolin G, Patrizi G, Cappelli S, Villani GQ, Piepoli M, Zobbi G, Nicosia E, Ardissino D. ALLiance for sEcondary PREvention after an acute coronary syndrome. The ALLEPRE trial: A multicenter fully nurse-coordinated intensive intervention program. Am Heart J. 2018 Sep;203:12-16. doi: 10.1016/j.ahj.2018.06.001. Epub 2018 Jun 12. PMID 29966801
- [Background] Buckley BJR, de Koning IA, Harrison SL, Fazio-Eynullayeva E, Underhill P, Kemps HMC, Lip GYH, Thijssen DHJ. Exercise-based cardiac rehabilitation vs. percutaneous coronary intervention for chronic coronary syndrome: impact on morbidity and mortality. Eur J Prev Cardiol. 2022 May 25;29(7):1074-1080. doi: 10.1093/eurjpc/zwab191. PMID 34788451